CLINICAL TRIAL: NCT06076278
Title: Effects of Home Based Resistance Training as Compared to Supervised Resistance Training Exercise in the Management of Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUI/CTR/2023/17
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive home based resistant training and the second will receive clinic based resistant training. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Resistant Training) (Active Comparator): Patients in this group will recieve Clinic based resistant training . A total of 12 sessions will be conducted over a period of 4 week 3 days a week.
  Interventions: Procedure: resistance exercise
- Group B (Home Based resistant training) (Experimental): Patients will recieve home based resistant training. A total of 12 sessions will be conducted over a period of 4 week ,3 days a week .
  Interventions: Procedure: resistance exercise

INTERVENTIONS:
Procedure: resistance exercise — Isometrics contraction of quadriceps Supine straight leg raise Leg lifts in prone position Passive knee flexion Passive knee extension Resistance knee extension Resistance knee flexion Isometric terminal knee extension in lying and mini-squat Concentric and isometric knee extension and flexion in sitting Frequency: A total of 12 sessions, thrice a week, for 4 consecutive weeks. Time Duration: Approx. 25 to 30minutes

SUMMARY:
Knee osteoarthritis is a degenerative pathology that is characterized by structural changes in the joint, such as joint space narrowing, thickening of the joint capsule, and cartilage degeneration that encourages friction between the bone surfaces and causes pain, which is thought to be a major symptom of knee osteoarthritis. Knee osteoarthritis (OA) treatment focuses on reducing pain while also enhancing function and quality of life by resistant training and Home-based exercise, a time-effective and practical treatment option for people with chronic conditions. As the past literature states that home based trainings are cost and time effective, However there is deficient evidence regarding effectiveness of home based strength training in case of knee osteoarthritis. More evidence is therefore needed in this regard.

DETAILED DESCRIPTION:
As the investigators know knee osteoarthritis (KOA) is common in elderly people, causes pain, loss of physical functioning, and disability. Knee osteoarthritis (OA) treatment focuses on reducing pain while also enhancing function and quality of life. Increased interest in non-pharmacologic treatments for OA is a result of declining enthusiasm for cyclooxygenase-2 inhibitors as a means of treating knee OA pain and failing clinical trials of OA medications that aim to change the illness. The two hallmarks of non-pharmacologic treatment are resistance training (RT) exercise programs and educational self-management (SM) programs and It has been evident in recent years that RT can have a favorable impact on activity-related energy expenditure, total free-living energy expenditure, and resting energy expenditure (REE) (AEE).Home based training; Home-based exercise, a time-effective and practical treatment option for people with chronic conditions like KOA, is becoming more valued by rehabilitation professionals and researchers. It can performed by patients individually at home, The goal of home-based and hospital-based exercise is the same; that is, to relieve pain and improve function by strengthening lower limb muscles, improving neuromuscular control, and range of joint motion in the affected knees. The main aim of the study is to determine the effectiveness of home-based resistance training as compared to supervised resistance training exercises in the management of knee osteoarthritis in terms of pain, ROM , disability, muscle strength and spatiotemporal parameter of gait. The participants meeting the eligibility criteria will be recruited, followed by random allocation to 2 groups. Both groups will receive standard treatment protocol which consists resistant training .12 sessions will be provided on alternative days. Pre and Post assessment of will be noted .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 60 years experiencing knee pain.
* Both male and female.
* Patients with grade 1 to 3 OA based on Kellgren Lawrence classification of knee OA.
* Those participants with 4-8 on NPRS

Exclusion Criteria:

* Individuals with serious pathology such as malignancy, inflammatory disorder or infection.
* Individual with history of knee surgery or replacement.
* Those patients who have received physiotherapy from last 2 months.
* Those patients who have received any surgical treatment for SIJ dysfunction

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 4 week
  Pain will be measured using the Numeric Pain Rating Scale, which is an 11-item scale.The higher the score the greater will be pain severity
Disability level of participant | 4 weeks
  Disability will be assessed using Western Ontario and McMaster University Osteoarthritis Index. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations
Muscle strength | 4 weeks
  measured by using Modified Sphygmomanometer Dynamometry
Gait Cadence | 4 weeks
  Cadence (steps/min) = steps counted x 60/time (s)
Range of motion | 4 weeks
  Description measured by using Goniometer
Gait Stride length | 4 weeks
  Stride length (m) = speed (m/s) x cycle time (s)
Gait Speed | 4 weeks
  Gait Speed (m/s) = distance (m) / time (s)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan